CLINICAL TRIAL: NCT03030742
Title: Postpartum Opioid Prescribing Patterns and Patient Utilization
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Society for Maternal-Fetal Medicine (Unknown)
Responsible Party: Principal Investigator, Lynn M Yee, Assistant Professor, Northwestern University
Other Study IDs: NortherwesternU
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Postpartum; Opioid Use; Post-operative; Cesarean Delivery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-cesarean delivery: Women who have undergone cesarean delivery
  Interventions: Other: Survey
- Post-vaginal delivery: Women who have undergone vaginal delivery
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A survey will be administered at two time points (time of hospital discharge and 2-4 weeks postpartum) to determine:
  * Satisfaction with pain control 2-4 weeks postpartum
  * Patient-reported use of opioid medication postpartum (receipt of prescription, filling of prescription, if refill was obtained, and number of opioid pills remaining at the time of follow-up)
  * Patient characteristics associated with high opioid use
  * Methods of storage and disposal of unused opioids
  Other Names: Survey/Questionnaire

SUMMARY:
This study seeks to investigate the prescribing patterns and patient utilization of opioid pain medication in the postpartum setting. Postpartum women will be surveyed prior to hospital discharge and again at 2-4 weeks postpartum in order to assess the number of opioid tablets they used (in relation to the number prescribed), pain satisfaction, and storage/disposal of any remaining opioid tablets.

DETAILED DESCRIPTION:
Opiate abuse is a national epidemic and has paralleled the increase in opioid prescriptions, with diversion of surplus medication playing a key contributing role. As the majority of reproductive age women in the U.S. will experience childbirth, understanding opioid prescription patterns and patient opioid utilization in the postpartum period is critical.

Postpartum women will be recruited during a 9-month period to take part in pre-hospital discharge and 2-4 week postpartum surveys to prospectively assess opioid medication use with regard to quantity of opioid tablets prescribed and quantity used, storage and disposal of unused opioids and satisfaction with pain control.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver during the recruitment period
* English-speaking
* Opiate-naïve (as determined by admission medication reconciliation)
* Receive oral opioid medications during inpatient postpartum admission
* 18 years or older

Exclusion Criteria:

* Contraindication to NSAID use
* Required use of general anesthesia without concurrent neuraxial analgesia
* Undergo hysterectomy, or unanticipated surgical procedures during the postpartum period
* Are admitted to the intensive care unit during their admission.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women who are postpartum
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Postpartum outpatient opioid use | 8 weeks
  Self reported number of opioid tablets used at time of postpartum survey administered 2-4 weeks postpartum

SECONDARY OUTCOMES:
Satisfaction with outpatient pain control | 8 weeks from time of hospital discharge
  Satisfaction with pain control at the time of postpartum survey administered 2-4 weeks postpartum
Proper disposal/storage of remaining opioid tablets | 8 weeks from time of discharge
  Proportion of patients who report proper disposal/storage of remaining opioid tablets at the time of postpartum survey administered 2-4 weeks postpartum
High opioid use | 8 weeks from time of hospital discharge
  Comparison of characteristics of women with >50% remaining versus <50% remaining of prescribed opioid tablets

CONTACTS AND LOCATIONS:
Overall Officials: Nevert Badreldin, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers and other drugs among women--United States, 1999-2010. MMWR Morb Mortal Wkly Rep. 2013 Jul 5;62(26):537-42. PMID 23820967
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Pfuntner A, Wier LM, Stocks C. Most Frequent Procedures Performed in U.S. Hospitals, 2010. 2013 Feb. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #149. Available from http://www.ncbi.nlm.nih.gov/books/NBK132428/ PMID 23596641
- [Background] Peirce GL, Smith MJ, Abate MA, Halverson J. Doctor and pharmacy shopping for controlled substances. Med Care. 2012 Jun;50(6):494-500. doi: 10.1097/MLR.0b013e31824ebd81. PMID 22410408
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Paulozzi LJ, Mack KA, Hockenberry JM; Division of Unintentional Injury Prevention, National Center for Injury Prevention and Control, CDC. Vital signs: variation among States in prescribing of opioid pain relievers and benzodiazepines - United States, 2012. MMWR Morb Mortal Wkly Rep. 2014 Jul 4;63(26):563-8. PMID 24990489
- [Background] Mkontwana N, Novikova N. Oral analgesia for relieving post-caesarean pain. Cochrane Database Syst Rev. 2015 Mar 29;2015(3):CD010450. doi: 10.1002/14651858.CD010450.pub2. PMID 25821010
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Sun EC, Darnall BD, Baker LC, Mackey S. Incidence of and Risk Factors for Chronic Opioid Use Among Opioid-Naive Patients in the Postoperative Period. JAMA Intern Med. 2016 Sep 1;176(9):1286-93. doi: 10.1001/jamainternmed.2016.3298. PMID 27400458
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844